CLINICAL TRIAL: NCT00637039
Title: A Phase 1, Open-label, Multiple-dose, Dose Escalation Study to Assess the Safety, Tolerability and Pharmacokinetics of AZD8931 in Patients With Advanced Solid Malignancies
Brief Title: Study of AZD8931 in Patients With Advanced Solid Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D0102C00002; AZD8931 Study 002
Record Dates: First submitted 2008-03-10; First posted 2008-03-17 (Estimated); Last update posted 2013-03-12 (Estimated); Status verified 2013-03

CONDITIONS: Advanced Solid Malignancies
Keywords: Advanced cancer; Solid tumour; Solid malignancies; Neoplasms
MeSH Terms: conditions — Neoplasms | interventions — AZD 8931

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: AZD8931 — Tolerability and Pharmacokinetics of AZD8931 in Patients with Advanced Solid Malignancies.

SUMMARY:
The main purpose of this study is to explore the safety and tolerability of multiple ascending doses (MAD) of AZD8931 in patients with advanced solid malignancies

ELIGIBILITY:
Inclusion Criteria:

* Cancer which is refractory to standard therapies, or for which no standard therapies exist. Inclusion is irrespective of stage of disease or extent of prior therapy.
* Histologically or cytologically confirmed solid, malignant tumour.

Exclusion Criteria:

* Receipt of any of the following treatments within 4 weeks prior to study entry: chemotherapy (within 6 weeks for nitrosurea or mitomycin C), radiotherapy, hormone therapy (except for androgen-deprivation therapy for patients with prostate cancer), immunotherapy and any other anti-cancer therapies.
* Unresolved toxicity (other than stable toxicity) from previous anti-cancer therapy, except alopecia.
* History of documented cardiac failure, angina pectoris requiring antianginal medication, evidence of transmural infarction on ECG, poorly controlled hypertension (systolic >180 mmHg or diastolic >100 mmHg), significant valvular disease or history of high risk dysrrhythmia (such as ventricular fibrillation or ventricular tachycardia [includes ventricular triplets]).
* Resting ECG with measurable QTc interval of > 460 msec at 2 or more time-points within a 24-hour time period, or history of prolonged QTc syndrome.
* The presence of any ocular disease or condition that is active or is likely to flare up during the course of the study or any systemic disease/condition that is affecting or has affected the eye in the past and may flare up, or the treatment of which may have an adverse effect on the eye. Eye conditions that are stable and of long standing, such as scars from trauma, pinguecula, atrophic pterygia etc, should not be considered as reasons to exclude the patient.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2008-02; Primary Completion 2009-06 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Explore the safety and tolerability of multiple ascending doses (MAD) of AZD8931 in patients with advanced solid malignancies, by assessment of AEs, lab findings, physical examinations, vital signs, cardiac monitoring and ophthalmological examinations

SECONDARY OUTCOMES:
To identify the maximum tolerated dose (MTD) of AZD8931 following repeated twice daily administration, by assessment of dose limiting toxicities (DLT)
To explore the pharmacokinetics (PK) of single doses of AZD8931 in patients with advanced solid malignancies
To explore the pharmacokinetics (PK) of multiple doses of AZD8931 in patients with advanced solid malignancies

CONTACTS AND LOCATIONS:
Overall Officials: S. Tjulandin, Principal Investigator — GU Russian Oncology Research Centre; Serban Ghiorghiu, Study Director — AstraZeneca
Locations (3):
- Research Site, Berlin, Germany
- Russia (2):
  - Research Site, Moscow
  - Research Site, Saint Petersburg

REFERENCES:
- [Derived] Tjulandin S, Moiseyenko V, Semiglazov V, Manikhas G, Learoyd M, Saunders A, Stuart M, Keilholz U. Phase I, dose-finding study of AZD8931, an inhibitor of EGFR (erbB1), HER2 (erbB2) and HER3 (erbB3) signaling, in patients with advanced solid tumors. Invest New Drugs. 2014 Feb;32(1):145-53. doi: 10.1007/s10637-013-9963-6. Epub 2013 Apr 16. PMID 23589215